CLINICAL TRIAL: NCT00374933
Title: Non-Myeloablative Conditioning With Allogeneic Peripheral Blood Progenitor Cell Transplantation Followed by Prophylactic Activated Donor Lymphocyte Infusion (DLI) for the Treatment of High Risk Acute Leukemia/MDS
Brief Title: Enhancing Graft vs Leukemia Via Delayed Ex-Vivo Co-Stimulated DLI After Non-Myeloablative Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 08405
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
Keywords: AML; ALL; MDS; Allogeneic transplant; Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome; Adoptive cell therapy; Non-myeloablative
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes

ARMS (1):
- 1 (Experimental): "Prophylactic" delayed activated donor lymphocyte infusion (ADLI) after non-myeloablative conditioning and allogeneic peripheral blood cell stem cell transplantation
  Interventions: Drug: Non-myeloablative allogeneic stem cell transplant with prophylactic activated DLI; Drug: "Prophylactic" delayed ADLI; Drug: "Prophylactic" delayed activated donor lymphocyte infusion

INTERVENTIONS:
Drug: Non-myeloablative allogeneic stem cell transplant with prophylactic activated DLI — "Prophylactic" delayed activated donor lymphocyte infusion (ADLI) after non-myeloablative conditioning and allogeneic peripheral blood cell stem cell transplantation
Drug: "Prophylactic" delayed ADLI — "Prophylactic" ADLI after non-myeloablative conditioning and allogeneic peripheral blood cell stem cell transplantation
Drug: "Prophylactic" delayed activated donor lymphocyte infusion — "Prophylactic" delayed activated donor lymphocyte infusion (ADLI) after non-myeloablative conditioning and allogeneic peripheral blood cell stem cell transplantation

SUMMARY:
This is a new platform in non-myeloablative allogeneic stem cell transplantation to improve survival by harnessing the immunologic potential of donor T-cells to induce and maintain long-term remissions in patients with hematologic malignancies without undue toxicity. This study involves is the first study in humans directed at optimizing the graft vs leukemia effect by infusing activated T-cells from healthy donors prophylactically, months after recovery from the initial transplant. Investigators are studying whether the activation of donor cells prior to infusion will enhance the patient's ability to "seek and destroy" residual malignant cells while also helping the immune system to fight infection without increasing the immune reaction against the host.

ELIGIBILITY:
Patient-related Parameters:

* Patients must have a healthy histocompatible donor (A, B and DR match); either sibling or unrelated volunteer identified through the NMDP
* Age between 18 and 70 years old
* Life expectancy greater than 3 months.
* ECOG performance status 0-1.
* Patients must have acceptable organ function:
* total bilirubin <2.0
* AST and ALT < 3 x normal, unless increases are thought to be either from non-hepatic causes (i.e hemolysis) or related to underlying disease (such as liver involvement with leukemia);
* creatinine <2.0 or creatinine clearance >40 ml/min (calculated or collected);
* Cardiac: An ejection fraction >40% on MUGA or echocardiogram;
* Pulmonary: corrected DLCO >50%

Exclusion Criteria:

Subjects:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study. Patients must have recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients with uncontrolled or untreated central nervous system involvement
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV positive patients are excluded
* Pregnant women
* Patients who are breastfeeding

Donors:

* Sibling donors will be evaluated according to the standard practice of the University of Pennsylvania Bone Marrow and Stem Cell Transplant Program
* Unrelated donor evaluations and consent will be performed by an NMDP donor center according to standard guidelines and procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and feasibility of administering prophylactic donor lymphocyte infusion (DLI) after non-myeloablative transplant (NMT). | Six months after last patient entered on study.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Goldstein, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States